CLINICAL TRIAL: NCT04261686
Title: A Prospective, Multi-Center, Non-Randomized Clinical Study of the BARD® COVERA Arteriovenous (AV) Stent Graft in the Treatment of Stenosis in the Venous Outflow of AV Fistula Access Circuits (AVeNEW) Post Approval Study
Brief Title: Post Approval Study of the BARD® COVERA™ Arteriovenous (AV) Stent Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDPI-19-001
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- COVERA Vascular Covered Stent (Other): COVERA Vascular Covered Stent for the treatment of stenotic lesions in the upper extremity venous outflow of the arteriovenous (AV) access circuit of hemodialysis subjects dialyzing with an AV fistula.
  Interventions: Device: Covera Vascular Covered Stent

INTERVENTIONS:
Device: Covera Vascular Covered Stent — This is a single-arm study. All subjects will receive the Covera Vascular Covered Stent

SUMMARY:
The objective of this study is to collect post-market, real-world safety and effectiveness data of the COVERA Vascular Covered Stent for the treatment of stenotic lesions in the upper extremity venous outflow of the arteriovenous (AV) access circuit.

DETAILED DESCRIPTION:
Prospective, multi-center, non-randomized clinical study designed to assess the long-term safety and effectiveness of the COVERA Vascular Covered Stent for the treatment of stenotic lesions in the upper extremity venous outflow of the AV access circuit of hemodialysis subjects dialyzing with an arteriovenous (AV) fistula.

ELIGIBILITY:
Clinical Inclusion Criteria

1. Subject must voluntarily sign and date the Informed Consent Form (ICF) prior to collection of study data or performance of study procedures.
2. Subject must be either a male or non-pregnant female ≥ 21 years of age with an expected lifespan sufficient to allow for completion of all study procedures.
3. Subject must be willing to comply with the protocol requirements, including clinical and telephone follow-up.
4. Subject must have an upper extremity AV fistula that has undergone at least one successful dialysis session with two-needle cannulation, prior to the index procedure.
5. Subject must have angiographic evidence of a stenosis ≥ 50% (by visual estimation) located in the venous outflow of the AV access circuit and present with clinical or hemodynamic evidence of AV fistula dysfunction.
6. The target lesion must be ≤ 9cm in length. Note: multiple stenoses may exist within the target lesion.
7. The reference vessel diameter of the adjacent non-stenotic vein must be between 5.0 and 9.0mm.

Exclusion Criteria:

Clinical Exclusion Criteria

1. The subject is dialyzing with an AV graft.
2. The target lesion has had a corresponding thrombosis treated within 7 days prior to the index procedure.
3. The hemodialysis access is located in the lower extremity.
4. The subject has an infected AV fistula or uncontrolled systemic infection.
5. The subject has a known uncontrolled blood coagulation/bleeding disorder.
6. The subject has a known allergy or hypersensitivity to contrast media which cannot be adequately pre-medicated.
7. The subject has a known hypersensitivity to nickel-titanium (Nitinol) or tantalum.
8. The subject has another medical condition, which, in the opinion of the Investigator, may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures and follow-up.
9. The subject is currently participating in an investigational drug or another device study that has not completed the study treatment or that clinically interferes with the study endpoints. Note: Studies requiring extended follow-up visits for products that were investigational, but have since become commercially available, are not considered investigational studies.
10. Additional stenotic lesions (≥ 50%) in the venous outflow that are > 3cm from the edge of the target lesion and are not successfully treated (defined as ≤ 30% residual stenosis) prior to treating the target lesion.
11. An aneurysm or pseudoaneurysm is present within the target lesion.
12. The location of the target lesion would require the COVERATM Vascular Covered Stent be deployed across the elbow joint.
13. The target lesion is located within a stent.
14. The location of the target lesion would require that the COVERA™ Vascular Covered Stent be deployed at or across the segment of fistula utilized for dialysis needle puncture (i.e., "cannulation zone").
15. The location of the target lesion would require that the COVERA™ Vascular Covered Stent be placed in the central veins (subclavian, brachiocephalic, Superior Vena Cava (SVC)) or under the clavicle at the thoracic outlet.
16. There is incomplete expansion of an appropriately sized angioplasty balloon to its expected profile, in the operator's judgment, during primary angioplasty at the target lesion.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Safety through 30 days | Through 30 days following index procedure
  Freedom from any adverse event(s), localized or systemic, that reasonably suggest the involvement of the AV access circuit that require or result in any of the following alone or in combination: additional interventions, in-patient hospitalization or prolongation of an existing hospitalization; or death.
Target Lesion Primary Patency (TLPP) | 1, 3, 6, 12, 18, 24, and 36 months following post-index procedure
  The interval following the index intervention until the next clinically driven reintervention at or adjacent to the original treatment site, or until the extremity is abandoned for permanent access.
Access Circuit Primary Patency (ACPP) | 1, 3, 6, 12, 18, 24, and 36 months post index procedure
  The interval following the index intervention until the next access thrombosis or repeated intervention.
Rate of Device and Procedure Related Adverse Events involving the access circuit | 1, 3, 6, 12, 18, 24, and 36 months post index procedure.
  Rate of device and procedure related adverse events (AEs) involving the access circuit.
Total Number of Arteriovenous (AV) Access Circuit Reinterventions | 1, 3, 6, 12, 18, 24, and 36 months post index procedure
  Number of reinterventions to the arteriovenous (AV) access circuit until access abandonment or through study completion.
Total Number of Target Lesion Reinterventions | 1, 3, 6, 12, 18, 24, and 36 months post index procedure
  Number of reinterventions to maintain target lesion patency
Index of Patency Function (IPF) | 1, 3, 6, 12, 18, 24, and 36 months post index procedure
  Time from the index study procedure to study completion or access abandonment divided by the number of visits for a reintervention performed on the arteriovenous (AV) access circuit in order to maintain vascular access for hemodialysis.
Index of Patency Function for Target Lesion | 1, 3, 6, 12, 18, 24, and 36 months post index procedure
  Time from the index study procedure to study completion or complete access abandonment divided by the number of visits for a reintervention performed at the target lesion in order to maintain vascular access for hemodialysis.
Post-Intervention Secondary Patency | 1, 3, 6, 12, 18, 24, and 36 months post index procedure
  The interval after the index intervention until the access is abandoned.
Acute Technical Success for Stent Graft Placement | At time of index procedure
  Defined as the successful deployment, based on the operator's opinion, of the implant to the intended location assessed at the time of the index procedure.
Acute Procedural Success | At time of index procedure
  Defined as anatomic success and resolution of the pre-procedural clinical indicator(s) (clinical success) of a hemodynamically significant stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Bart Dolmatch, M.D., Principal Investigator — The Palo Alto Medical Foundation
Locations (11):
- United States (11):
  - Arizona Kidney Disease and Hypertension Center Medical Research Services, Phoenix, Arizona
  - Yale University, New Haven, Connecticut
  - Chicago Access Care, Westmont, Illinois
  - Kidney Care & Transplant Services of New England, West Springfield, Massachusetts
  - Michigan Vascular Center, Flint, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Minnesota Vascular and Surgery Center, New Brighton, Minnesota
  - North Carolina Nephrology, Raleigh, North Carolina
  - Providence Access Care, Providence, Rhode Island
  - Dallas Renal Group, Dallas, Texas
  - San Antonio Kidney and Disease Access Center, San Antonio, Texas

REFERENCES:
- [Derived] Dolmatch B, Saber T, Underwood M; and AVeNEW PAS trial investigators. Six-Month Outcomes from the Prospective, Multi-Center, Non-Randomized Clinical Study of the COVERA() Arterio VeNous (AV) Stent Graft in the Treatment of Stenosis in the VEnous OutfloW of AV Fistula Access Circuits (AVeNEW PAS). Cardiovasc Intervent Radiol. 2025 Apr;48(4):460-471. doi: 10.1007/s00270-024-03930-7. Epub 2025 Jan 9. PMID 39789255